CLINICAL TRIAL: NCT01501383
Title: A Phase 2b, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Dose-Ranging Study to Evaluate the Efficacy and Safety of VX-765 in Subjects With Treatment-Resistant Partial Epilepsy With a 24-Week Open-Label Extension
Brief Title: A Study to Evaluate the Efficacy and Safety of VX-765 in Subjects With Treatment-Resistant Partial Epilepsy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated by Sponsor
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VX11-765-402
Record Dates: First submitted 2011-12-15; First posted 2011-12-29 (Estimated); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- VX-765 Dose 1 Part A (Active Comparator)
  Interventions: Drug: VX-765 Part A
- VX-765 Dose 2 Part A (Active Comparator)
  Interventions: Drug: VX-765 Part A
- VX-765 Dose 3 Part A (Active Comparator)
  Interventions: Drug: VX-765 Part A
- VX-765 Dose 4 Part A (Active Comparator)
  Interventions: Drug: VX-765 Part A
- Placebo Dose Part A (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- VX-765 Dose Part B (Active Comparator)
  Interventions: Drug: VX-765 Part B

INTERVENTIONS:
Drug: VX-765 Part A — Tablets of VX-765 given at different doses based on treatment group in Part A
  Arms: VX-765 Dose 1 Part A; VX-765 Dose 2 Part A; VX-765 Dose 3 Part A; VX-765 Dose 4 Part A
Drug: Placebo — Matching placebo
  Arms: Placebo Dose Part A
Drug: VX-765 Part B — Tablets of VX-765 given at different doses based on patients who meet the study eligibility criteria for Part B
  Arms: VX-765 Dose Part B

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety and tolerability of VX-765 in subjects with treatment-resistant partial epilepsy.

ELIGIBILITY:
Part A and Part B Inclusion Criteria:

* Males or females aged 18 to 64 years with a body mass index between 18 and 35 (kg/m2)
* Subjects who have completed the assigned study treatment in Part A may enter Part B if eligible per protocol
* Male or female subjects must agree to use acceptable contraceptive methods, as described in the protocol
* Must have a diagnosis and history of treatment-resistant partial-onset epilepsy for which they are taking 1 to 4 concomitant AEDs at the time of Screening Period
* Have had at least 1 electroencephalogram consistent with partial epilepsy
* Must have had at least 6 partial-onset seizures and a seizure-free period of no more than 3 weeks (21 days) during the Baseline Period.
* Subjects with stable medical conditions (e.g., cannot have a condition that will interfere with the conduct of the study or cause a known increase in risk of the intervention) as determined by the principal investigator
* Must be able and willing to provide written informed consent to participate
* Must be able to understand and comply with protocol requirements and instructions

Part A and Part B Exclusion Criteria:

* Subjects who are male and their female partner (if of childbearing potential) does not agree to use medically approved methods of contraception as described in the protocol for the duration od the study and for 90 days after last dose of study drug
* Subjects who are male and have a female partner who is pregnant, nursing, or is planning to become pregnant during the study period, or within 90 days of the last dose of study drug.
* Subjects who are pregnant or lactating, or who are of reproductive potential who do not agree to use medically approved birth control methods
* History of nonepileptic, transient alterations in consciousness
* History of status epilepticus in the past 12 months before the screening visit
* Subjects whose seizure frequency cannot be quantified (i.e. seizures with no discrete beginning or end, or period between seizures)
* Subjects who have a significant medical illness including kidney, liver, pulmonary, or gastrointestinal disease; or unstable or poorly controlled conditions such as hypertension, diabetes, or angina pectoris, as judged by the investigator.
* Have a clinically significant psychiatric illness as judged by the investigator
* Subjects who have had an active suicidal plan/intent or active suicidal thoughts, or suicide attempt as defined in the protocol
* Clinically significant laboratory abnormalities during the Screening Visit/Baseline Period, as judged by the investigator
* Subjects who have had serious adverse events (SAEs) thought to be related to study drug that led to discontinuation during Part A may not participate in Part B
* Active hepatitis B, hepatitis C, or human immunodeficiency virus
* Positive drug screen at screening or during the Baseline Period (excluding any allowed prescribed medications) and/or a history of alcoholism or drug addiction within past 2 years
* Subjects on felbamate with fewer than 18 month of continuous felbamate exposure at the time of the Screening Visit or with significant adverse reactions to felbamate
* Subjects treated with vigabatrin fewer than 2 years prior to the Screening Visit or who have a prior history of treatment with vigabatrin without a documented stable examination by an ophthalmologist as defined in the protocol
* Using prohibited medications or treated with any systemic immunosuppressant
* Have experienced a symptomatic viral, fungal, or bacterial infection requiring systemic treatment within 7 days prior to the first dose of study drug
* A current or prior history of illness precluding them from immunomodulatory therapy (e.g., history of recurrent infections)
* Have donated any blood or have had a significant loss of blood (500 mL) as defined in the protocol
* Have participated in any other clinical studies involving an investigational product or device and have received the last dose of the study drug associated with that clinical study within 30 days or 5 half-lives (whichever is longer) of the Screening Visit
* Have participated in earlier VX-765 clinical studies and received at least one dose of study drug
* Subjects who have no completed the full 13-week Treatment Period in part A may not participate in Part B
* Any subject judged by the investigator, sponsor or designee to be inappropriate for the study

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2011-12; Primary Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Percent reduction in weekly seizure frequency during the Part A Late Treatment Period compared to the Part A Baseline Period | Up to 25 Weeks
Percent of subjects with 50% or greater reduction in weekly seizure frequency (responder-rate) during the Part A Late Treatment Period compared to the Part A Baseline Period | Up to 25 Weeks
Safety and tolerability as assessed by vital signs, standard 12-lead electrocardiograms (ECGs), laboratory assessments (serum chemistry, hematology, and urinalysis), and adverse events | Up to 56 Weeks
Safety and tolerability as determined by vital signs, standard 12-lead electrocardiograms (ECGs), laboratory assessments (serum chemistry, hematology, and urinalysis) and adverse events | Up to 56 Weeks

SECONDARY OUTCOMES:
Percent of subjects who are seizure-free during the Part A Late Treatment Period | Up to 25 Weeks
Percent reduction in seizure frequency during the entire Part A Treatment Period compared to the Part A Baseline Period | Up to 25 Weeks
Percent of subjects with 50% or greater reduction in seizure frequency (responder-rate) during the entire Part A Treatment Period compared to the Part A Baseline Period | Up to 25 Weeks
Percent of subjects who are seizure-free during the entire Part A Treatment Period | 13 Weeks
Maximum number of consecutive days that subjects do not have seizures at any time during the Part A Late Treatment Period | Up to 13 Weeks
Maximum number of consecutive days that subjects do not have seizures at any time during the entire Treatment Period | 13 Weeks
Pharmacokinetics (e.g AUC, Cmax) of VX-765, VRT-043198, and concomitant antiepileptic drug (AED) levels in blood | Up to 21 Weeks
Percent reduction in weekly seizure frequency compared to the Part A Baseline Period | Up to 56 Weeks
Percent of subjects with 50% or greater reduction in weekly seizure frequency (50% responder-rate) during the entire Part B Treatment Period compared to the Part A Baseline Period | Up to 56 Weeks
Percent of subjects with 75% or greater reduction in weekly seizure frequency (75% responder-rate) during the entire Part B Treatment Period compared to the Part A Baseline Period | Up to 56 Weeks
Percent of subjects who are seizure-free during the entire Part B Treatment Period | Up to 28 Weeks
Maximum number of consecutive days that subjects do not have seizures at any time during the entire Part B Treatment Period | Up to 28 Weeks
Percent increase in weekly seizure-free days compared to the Part A Baseline Period | Up to 56 Weeks

CONTACTS AND LOCATIONS:
Locations (24):
- United States (22):
  - Alabama, Northport, Alabama
  - Arizona, Phoenix, Arizona
  - Arizon, Phoenix, Arizona
  - Arkansas, Little Rock, Arkansas
  - California, Loma Linda, California
  - Florida, Bradenton, Florida
  - Florida, Wellington, Florida
  - Idaho, Boise, Idaho
  - Maryland, Baltimore, Maryland
  - Michigan, Farmington Hills, Michigan
  - Minnesota, Saint Paul, Minnesota
  - New York, New York, New York
  - New York, The Bronx, New York
  - North Carolina, Asheville, North Carolina
  - North Carolina, Charlotte, North Carolina
  - Ohio, Columbus, Ohio
  - Oklahoma, Oklahoma City, Oklahoma
  - Pennsylvania, Philadelphia, Pennsylvania
  - Texas, Dallas, Texas
  - Utah, Orem, Utah
  - Virginia, Charlottesville, Virginia
  - Washington, Renton, Washington
- Germany (2):
  - Germany, Bonn
  - Germany, Kork